CLINICAL TRIAL: NCT00565279
Title: Efficacy and Safety of ASF 1057 Cream 0.5% in the Treatment of Seborrhoeic Dermatitis: A Phase III Randomised, Double-Blind, Vehicle and Placebo Controlled, Parallel Groups, Multi-Centre Trial.
Brief Title: Efficacy and Safety of ASF1057 in the Treatment of Seborrhoeic Dermatitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astion Pharma A/S (Industry)
Responsible Party: Dr Peder Andersen, Astion Pharma A/S
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ASF1057-301
Record Dates: First submitted 2007-11-28; First posted 2007-11-29 (Estimated); Last update posted 2008-06-03 (Estimated); Status verified 2008-06

CONDITIONS: Seborrheic Dermatitis
Keywords: Seborrhoeic dermatitis
MeSH Terms: conditions — Dermatitis, Seborrheic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- ASF1057 (Experimental)
  Interventions: Drug: ASF1057
- ASF1057 placebo (Placebo Comparator)
  Interventions: Drug: ASF1057
- ASF1057 Vehicle (Placebo Comparator)
  Interventions: Drug: ASF1057

INTERVENTIONS:
Drug: ASF1057 — Twice daily, topical
Drug: ASF1057 — Twice daily, Topical
  Arms: ASF1057; ASF1057 placebo

SUMMARY:
A growing body of evidence supports the hypothesis that the pathophysiology of seborrhoeic dermatitis has a potentially causative neurogenic inflammatory aspect. ASF1057 is a new drug that acts through a modulation of neurogenic inflammation through important complementary mechanisms of action. This study will test the efficacy and safety of ASF1057 in the treatment of patients with seborrhoeic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate to severe seborrhoeic dermatitis

Exclusion Criteria:

* Other active skin diseases
* Use of certain systemic and topical treatments
* Extensive sun exposure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-05 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Proportion of responders, defined as patients with OSS ≤ 1 score units. | Baseline, day 7, day 14, and day 21

CONTACTS AND LOCATIONS:
Overall Officials: Peder M Andersen, MD, Study Director — Astion Pharma A/S